CLINICAL TRIAL: NCT05891327
Title: Effects of Lepidium Meyenii (Maca) Extract Supplementation on Male Sexual Funtion
Brief Title: Maca Extract in Sexual Dysfunction Male
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202303063
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-05

CONDITIONS: Sexual Dysfunction Male
MeSH Terms: interventions — MacA protein, E coli

STUDY DESIGN:
Intervention Model Description: assign 60 participants into the experimental group (n = 30) or placebo group (n = 30)
Who Masked: Participant, Investigator
Masking Description: A double-blind, matched-pair study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maca group (Experimental)
  Interventions: Dietary Supplement: Maca
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Maca — 2.25 g Lepidium meyenii (Maca) extract twice per day for 12 weeks
  Arms: Maca group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The purpose of this study was to investigate the effects of Lepidium meyenii (Maca) extract supplementation on male sexual funtion.

DETAILED DESCRIPTION:
All participants performed anthropometric measurements, blood collection and questionnaire survey at 0-week. A random, double-blind design will be used to assign 60 participants into the experimental group (n = 30) or placebo group (n = 30). All participants consumed either 2.25 g Lepidium meyenii (Maca) extract twice per day for 12 weeks. The anthropometric measurements, blood samples, and questionnaire survey were collected again at 6-week, 12-week, 16-week, and 24-week. Data will be analyzed by two-way mixed design ANOVA.

ELIGIBILITY:
Inclusion Criteria:

1. evaluated as sexual dysfunction for more than three months by physician
2. international index of erectile function (IIEF) score is less than or equal to 21
3. erectile hardness score (EHS) score is less than or equal to 3
4. aged over 18 years old

Exclusion Criteria:

1. unable to cooperate with the course of the treatment
2. suffering from sexually transmitted diseases such as Syphilis, AIDS and HPVs
3. had Radical Prostatectomy (total removal of the prostate gland)
4. suffering from active tumors in the prostate or pelvic area
5. suffering from Hypogonadism
6. anatomical deformation of the penis
7. men with penile prosthesis
8. suffering from psychotic disorder (manic disorder, chronic depression, etc.)
9. suffering from neurological diseases (multiple sclerosis, brain or spinal cord injuries, etc.)
10. using Permanent pacemaker
11. considered unsuitable to participate in this experiment according to the doctor
12. alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
IIEF-5 score | Baseline (before supplementation)
IIEF-5 score | 6 weeks of supplementation
IIEF-5 score | 12 weeks of supplementation
IIEF-5 score | 18 weeks of supplementation
IIEF-5 score | 24 weeks of supplementation
EHS score | Baseline (before supplementation)
EHS score | 6 weeks of supplementation
EHS score | 12 weeks of supplementation
EHS score | 18 weeks of supplementation
EHS score | 24 weeks of supplementation
level of PSA | Baseline (before supplementation)
level of PSA | 6 weeks of supplementation
level of PSA | 12 weeks of supplementation
level of PSA | 18 weeks of supplementation
level of PSA | 24 weeks of supplementation
Testosterone level | Baseline (before supplementation)
Testosterone level | 6 weeks of supplementation
Testosterone level | 12 weeks of supplementation
Testosterone level | 18 weeks of supplementation
Testosterone level | 24 weeks of supplementation
LH level | Baseline (before supplementation)
LH level | 6 weeks of supplementation
LH level | 12 weeks of supplementation
LH level | 18 weeks of supplementation
LH level | 24 weeks of supplementation
Level of FSH | Baseline (before supplementation)
Level of FSH | 6 weeks of supplementation
Level of FSH | 12 weeks of supplementation
Level of FSH | 18 weeks of supplementation
Level of FSH | 24 weeks of supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan